CLINICAL TRIAL: NCT00962455
Title: Feedback Reports and E-learning to Support Spirometry Test Performance in Dutch Family Practices
Brief Title: Feedback Reports and e-Learning in Primary Care Spirometry
Acronym: FRESCO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Quartz Transmural Centre for the Helmond Region (Unknown); Elkerliek Hospital (Other)
Responsible Party: Tjard Schermer, senior researcher, Radboud University Nijmegen MC, Dept of Primary and Community Care
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UMCN-CARA-0001113
Record Dates: First submitted 2009-08-17; First posted 2009-08-20 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Respiratory Tract Diseases; Pulmonary Disease, Chronic Obstructive; Asthma
Keywords: Spirometry; Family Practice; Randomized Controlled Trial; Feedback; Intervention Studies
MeSH Terms: conditions — Respiratory Tract Diseases; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- e-learning & performance feedback (Experimental): Initial e-learning by studying CD-Rom 'Spirometry Fundamentals', followed by repeated periodic performance feedback on spirometry test quality
  Interventions: Other: e-learning & performance feedback
- Usual practice (Active Comparator): Usual practice regarding spirometry execution in family practice
  Interventions: Other: usual practice

INTERVENTIONS:
Other: e-learning & performance feedback — Initial e-learning by studying CD-Rom 'Spirometry Fundamentals', followed by repeated periodic performance feedback on spirometry test quality
  Arms: e-learning & performance feedback
Other: usual practice — Usual practice regarding spirometry execution in family practice
  Arms: Usual practice

SUMMARY:
Spirometry is a biomedical test to measure lung function in subject who (may) have a chronic respiratory condition. Performing the test requires a certain level of training and experience from the health care professional who conducts the test, and sufficient cooperation of the patient. Although the test is widely used in primary care in many countries, the quality of the test performance seems limited and needs improvement in order to avoid false-positive and false-negative test interpretations. In this study, the researchers investigated whether a combination of e-learning and bimonthly written performance feedback to family practice nurses and assistance regarding their spirometry tests improves the rate of adequate tests.

ELIGIBILITY:
Inclusion Criteria for Family Practices:

* collaboration with Elkerliek Hospital Helmond through regional integrated care support service ('QUARTZ')
* purchased spirometer through this support service
* have implemented spirometry as a part of routine patient care

Inclusion Criteria for Patients:

* registered in one of the participating family practices
* performed a spirometry test as a part of routine care during the observation period of the study

Exclusion Criteria for Patients:

* age < 10 years

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1135 (Actual)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Proportion of spirometry tests with ≥2 acceptable blows according to 2005 ERS/ATS criteria that were also repeatable for both FEV1 and FVC | 12 months prospective follow-up

SECONDARY OUTCOMES:
Proportions of tests with ≥2 acceptable blows according to 2005 ERS/ATS criteria | 12 months prospective follow-up
Proportions of spirometry tests with ≥2 blows meeting 2005 ERS/ATS end-of-test criteria | 12 months prospective follow-up
Proportions of spirometry tests with A to C grade according to scholastic-type quality grading system by Ferguson et al (2000) | 12 months prospective follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Tjard R Schermer, PhD, Principal Investigator — Radboud University Medical Center; Alan J Crockett, PhD, Principal Investigator — The University of Adelaide; Willem Pieters, MD, PhD, Principal Investigator — Elkerliek Hospital
Locations (1):
- Radboud University Nijmegen Medical Centre, Department of Primary and Community Care, Nijmegen, Netherlands